CLINICAL TRIAL: NCT07132138
Title: Scooter Board Activities Versus Core Stability Exercises on Enhancing Trunk Postural Control and Balance in Children With Diplegic Cerebral Palsy: A Randomized Comparative Trial
Brief Title: Scooter Board Activities Versus Core Stability Exercises
Acronym: CP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Omnya Samy Abdallah Ghoneim, Lecturer, Department of Physical Therapy for Woman and Pediatric Health, Faculty of Physical Therapy, King Salman International University (KSIU), Sharm El-sheikh, Egypt., King Salman International university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study 4
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diplegic Cerebral Palsy
Keywords: Scooter Board Activities; Core Stability Exercises; Trunk Postural Control; Balance; Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The selected subjects will be divided into two groups of equal numbers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scooter Board Activities (Experimental): Received a designed physical therapy program in addition to scooter board activities.
  Interventions: Other: Scooter Board Activities
- Core Stability Exercises (Active Comparator): Received a designed physical therapy program in addition to core stability exercises.
  Interventions: Other: Core Stability Exercises

INTERVENTIONS:
Other: Scooter Board Activities — Scooter board bear walk. Scooter board crab walk. Sitting on scooter board, use it to move forward and backward, move the pool rings from one end to another.
  Cross sitting on scooter board, pulls along the rope using his/her hands Sit with knees pulled into the chest (like a bug pose) and move around with arms only.
  Prone over scooter board, pulling rope to move forward. Pull self along an anchored rope to retrieve items Scooter rolls outs. Place knees on floor and hands holding the edge of the front scooter board. Push board out a few inches then pull back, the further you roll, the harder it gets.
  8- Kneeling, Push self forward and backward with the use of a therapy ball (lots of Motor Planning).
  Supine flexion on scooter board, Clip clothespins to a rope hanging above.
  Other Names: Physical therapy program
  Arms: Scooter Board Activities
Other: Core Stability Exercises — Bridges Bird-dog Sit-ups on therapy ball Static and dynamic trunk holds
  Other Names: Physical therapy program
  Arms: Core Stability Exercises

SUMMARY:
Children with diplegic cerebral palsy (CP) often experience impaired trunk control and balance, which limits functional mobility. Core stability exercises are commonly used in pediatric physical therapy to improve trunk control. Scooter board activities, which challenge trunk stability through dynamic movement, may offer an engaging alternative. This study aims to compare the effects of these two interventions.

DETAILED DESCRIPTION:
Children with spastic diplegic cerebral palsy (CP) often present with impaired trunk postural control and reduced balance stability, which negatively affect their functional independence, gait, and participation in daily activities.

Core stability training is widely recognized in pediatric rehabilitation as a method to enhance trunk strength and improve postural alignment.

Scooter board activities, however, add an element of dynamic movement, sensory stimulation, and task-oriented play, potentially offering greater engagement and functional carryover.

This study directly compares the two approaches in order to establish evidence-based guidance for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. CP with a diplegia
2. Age 6 to 10 years
3. Grade 1 and 2 according to the Modified Ashworth scale (RW and Smith, 1987).
4. They could walk with limitation or holding on according to GMFCS (level I&II &III) (Palisano et al., 1997).
5. They were able to understand and follow verbal instructions

Exclusion Criteria:

1. Children with any surgical interference in the upper limb.
2. intellectual disability such that simple tasks could not be understood or executed.
3. Children with any visual or auditory problems.
4. Children with any surgical interference in the lower limb.
5. Children with any structural deformities in joints and bones of lower limbs.
6. Children who suffer from other diseases or associated disorders that interfered with physical activity

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | before and after 3 months of intervention
  The TCMS is a standardized observational assessment tool designed to evaluate static and dynamic trunk control in children with cerebral palsy (CP) during functional sitting tasks. It is particularly useful for detecting trunk impairments that affect balance, postural adjustments, and functional mobility.
  Scoring System
  Each item is scored 0-2:
  0 = Unable to perform or requires arm support/trunk compensation
  1. = Performs partially or with minimal compensations
  2. = Performs fully without compensations
  Total Score Range: 0-58
  Higher scores indicate better trunk control.

SECONDARY OUTCOMES:
Pediatric Balance Scale (PBS) | before and after 3 months of intervention
  The Pediatric Balance Scale is an adaptation of the Berg Balance Scale (BBS) specifically designed to assess functional balance in children. It evaluates both static and dynamic balance during everyday activities and is suitable for children with mild to moderate motor impairments, including those with cerebral palsy.
  Scoring System
  Each item scored on a 5-point ordinal scale (0-4):
  0 = Unable to perform
  1. = Needs maximal assistance or unable to complete safely
  2. = Needs moderate assistance or significant compensation
  3. = Performs independently but with mild instability or slowness
  4. = Performs independently and safely
  Total Score Range: 0-56
  Higher scores indicate better balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: Omnya samy, Lecturer, Principal Investigator — Badr University in Cairo, Egypt
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No